CLINICAL TRIAL: NCT06277115
Title: Acute, Intermediate and Long-term Effects of CPAP Therapy in Obstructive Sleep Apnoea: a Two-phase Interventional Trial.
Brief Title: Acute and Long-term Effects of CPAP in OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Esther Irene Schwarz, Deputy Clinical Director Department of Pulmonology, Principal Investigator, University of Zurich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BASEC Nr. 2020-02002
Record Dates: First submitted 2024-02-10; First posted 2024-02-26 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Obstructive Sleep Apnea of Adult
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Two-phase intervention: several weeks of CPAP therapy followed by two weeks CPAP therapy withdrawal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (therapy initiation followed by therapy withdrawal) (Other): Continuous positive airway pressure (CPAP)
  Interventions: Device: Continuous positive airway pressure (CPAP)

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP) — Nocturnal continuous positive airway pressure therapy is the gold standard treatment for symptomatic OSA. It provides positive pressure via a nasal or oronasal mask to prevent upper airway collapse during sleep.

SUMMARY:
Two-phase interventional non-inferiority trial (phase 1: at least 8 weeks of CPAP; phase 2: 2 weeks of CPAP withdrawal) including 32 patients with moderate to severe OSA to compare the physiological consequences of a short-term CPAP withdrawal to the changes in previously untreated OSA. The trial has been designed as a validation of the CPAP-withdrawal model. Baseline in-laboratory sleep studies will be performed prior to CPAP initiation, after 6-8 weeks on CPAP (treatment effect) and following 2 weeks of CPAP therapy withdrawal (withdrawal effect, effect of OSA recurrence).

DETAILED DESCRIPTION:
Background and Aim: Obstructive sleep apnoea (OSA) is a prevalent sleep-related breathing disorder. OSA is associated with daytime sleepiness, impaired quality of life, and adverse cardiovascular outcome. OSA can be effectively treated with nocturnal continuous positive airway pressure (CPAP) that restores normal breathing during sleep by preventing upper airway collapse. However, many patients in whom treatment of OSA is indicated are not able to adhere to CPAP, and the consequences of untreated OSA seem to differ between OSA phenotypes. Therefore, treatment alternatives to CPAP and a better understanding of treatment implications in different phenotypes of OSA are important targets in this research field. Thus, effective and controlled study designs are needed to address these research questions. Conventional randomised controlled CPAP trials are limited by low CPAP adherence resulting in an underestimation of the treatment effect. In addition, the impracticability of withholding an effective treatment from symptomatic patients resulting in inclusion of less symptomatic and patients with less severe OSA has limited the conclusions from previous trials. The CPAP therapy withdrawal model was introduced to allow studying the pathophysiological consequences of OSA and treatment effects of CPAP in an effective and controlled way. Optimally treated patients previously diagnosed with OSA established on CPAP therapy are included and undergo a short-term therapy interruption. A therapy withdrawal results in recurrence of OSA and pathophysiological changes can be attributed to OSA in this controlled model. However, it is uncertain whether the consequences of OSA during a short-term CPAP therapy withdrawal are comparable to long-term consequences of untreated OSA.

The aim of this two-phase interventional trial is to assess the effects of intermediate and long-term CPAP therapy as well as acute CPAP therapy withdrawal resulting in OSA recurrence compared to longstanding untreated OSA on cardiovascular and symptom outcomes in moderate and severe OSA. The objective is to study the comparability of conventional CPAP therapy trials with the CPAP withdrawal model in terms of evaluating relevant cardiovascular and patient-centred outcomes in OSA.

The investigators hypothesise that the treatment effect of CPAP in previously treatment-naïve patients with OSA - if adherent to CPAP - will support the same conclusions on OSA pathophysiology and therapy effects as a short-term CPAP withdrawal in treatment-adherent patients having a recurrence of OSA in response to CPAP withdrawal and thus support the use of this effective CPAP withdrawal model to use as future study design in interventional trials in OSA. It is hypothesised that the CPAP withdrawal is non-inferior to conventional CPAP trials in studying the effect on blood pressure and OSA-symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Untreated moderate or severe OSA with an apnoea-hypopnoea-index (AHI) of ≥ 20/h and an oxygen desaturation index (>3%-dips) of ≥ 20/h in an in-laboratory sleep study
* Epworth Sleepiness Scale Score ≥7/24 points
* Indication for CPAP therapy
* Written informed consent

Exclusion Criteria:

* Moderate or more severe obstructive or restrictive ventilatory disorder (FEV1 or FVC < 70%)
* Heart failure
* Other types of sleep-related breathing disorders, e.g. sleep-associated hypoventilation, central sleep apnoea, Cheyne Stoke's Breathing
* Hypoxic or hypercapnic respiratory failure (awake paO2 < 9 kPa or paCO2 > 6 kPa)
* Active treatment for OSA (CPAP, mandibular advancement device, hypoglossal nerve stimulation)
* Current professional driver or previous sleepiness-related accidents
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Nocturnal systolic blood pressure | at baseline and at 2 and at least 8 weeks of CPAP as well as after 1 and after 2 weeks of CPAP withdrawal
  Ambulatory blood pressure monitoring (ABPM)
Epworth Sleepines Scale Score (ESS) | at baseline and at 2 and at least 8 weeks of CPAP as well as after 1 and after 2 weeks of CPAP withdrawal
  Subjective sleepiness, ESS min-max 0-24 points and ESS >10 indicating pathological daytime sleepiness

SECONDARY OUTCOMES:
48h, 24h, diurnal and nocturnal systolic and diastolic blood pressure | at baseline and at 2 and at least 8 weeks of CPAP as well as after 1 and after 2 weeks of CPAP withdrawal
  ABPM
Office systolic and diastolic blood pressure | at baseline and at 2 and at least 8 weeks of CPAP as well as after 1 and after 2 weeks of CPAP withdrawal
  Morning office blood pressure
48h, 24h, diurnal, nocturnal and office heart rate | at baseline and at 2 and at least 8 weeks of CPAP as well as after 1 and after 2 weeks of CPAP withdrawal
  Heart rate from ABPM, office measurement and from sleep studies
Heart rate variability in the time and frequency domain (CV, RMSSD, pRR50, LF, HF, LF/HF) | at baseline and at 2 and at least 8 weeks of CPAP as well as after 1 and after 2 weeks of CPAP withdrawal
  Measures of heart rate variability (daytime and nighttime)
Blood pressure variability (BPV, systolic and diastolic) | at baseline and at 2 and at least 8 weeks of CPAP as well as after 1 and after 2 weeks of CPAP withdrawal
  BPV from ABPM and beat-to-beat blood pressure measurement
Baroreflex sensitivity (BRS) | at baseline and at 2 and at least 8 weeks of CPAP as well as after 1 and after 2 weeks of CPAP withdrawal
  Finometer
Arterial stiffness | at baseline and at 2 and at least 8 weeks of CPAP as well as after 1 and after 2 weeks of CPAP withdrawal
  ABPM
Measures of nocturnal hypoventilation (median and maximal transcutaneous partial pressure of CO2 = tcpCO2) | at baseline and at least 8 weeks of CPAP as well as after 2 weeks of CPAP withdrawal
  Sleep study parameters
Measures of nocturnal hypoxaemia (mean nocturnal oxygen saturation = ¢SpO2) | at baseline and at least 8 weeks of CPAP as well as after 2 weeks of CPAP withdrawal
  Sleep study parameters
Measures of nocturnal hypoxaemia (time spent with SpO2 below 90% = t<90) | at baseline and at least 8 weeks of CPAP as well as after 2 weeks of CPAP withdrawal
  Sleep study parameters
Measures of nocturnal hypoxaemia (hypoxic burden) | at baseline and at least 8 weeks of CPAP as well as after 2 weeks of CPAP withdrawal
  Sleep study parameters
Measures of OSA severity (apnoea-hypopnoea-index) | at baseline and at least 8 weeks of CPAP as well as after 2 weeks of CPAP withdrawal
  Sleep study parameters
Measures of OSA severity (oxygen-desaturation index) | at baseline and at least 8 weeks of CPAP as well as after 2 weeks of CPAP withdrawal
  Sleep study parameters
Sleepiness (Stanford Sleepiness Scale (SSS)) | at baseline and at 2 and at least 8 weeks of CPAP as well as after 1 and after 2 weeks of CPAP withdrawal
  Questionnaire; 7-point Likert scale to quantify a patient's sleepiness at the time the questionnaire is completed; highr scores indicate more sleepiness
Fatigue (fatigue severity scale (FSS)) | at baseline and at 2 and at least 8 weeks of CPAP as well as after 1 and after 2 weeks of CPAP withdrawal
  Questionnaire; 9 items, higher score indicates more fatigue
Disease-specific quality of life (Functional Outcomes of Sleep Questionnaire (FOSQ)) | at baseline and at 2 and at least 8 weeks of CPAP as well as after 1 and after 2 weeks of CPAP withdrawal
  Questionnaires, Disease-specific quality of life questionnaire to determine functional status in adults; measures are designed to assess the impact of disorders of excessive sleepiness on multiple activities of everyday living and the extent to which these abilities are improved by effective treatment; 30 items; higher scores are better
Superoxide dismutase | at baseline and at 2 and at least 8 weeks of CPAP as well as after 1 and after 2 weeks of CPAP withdrawal
  Marker of oxidative stress (U/ml)
Urinary catecholamines | at baseline and at 2 and at least 8 weeks of CPAP as well as after 1 and after 2 weeks of CPAP withdrawal
  Epinephrine and norepinephrine in morning urine (nnmol/mmol)
Pulse rise index (>6 beats per minute) | at baseline and at 2 and at least 8 weeks of CPAP as well as after 1 and after 2 weeks of CPAP withdrawal
  from nocturnal oximetry
Nocturnal oxymetry measures (¢SpO2, t<90, ODI-3%, ODI-4%) | at baseline and at 2 and at least 8 weeks of CPAP as well as after 1 and after 2 weeks of CPAP withdrawal
  nocturnal pulse oximetry

CONTACTS AND LOCATIONS:
Overall Officials: Esther I Schwarz, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland